CLINICAL TRIAL: NCT05951686
Title: The Effect of Two Different Anesthetic Methods on Gastrointestinal Motility in Patients Scheduled for Laparoscopic Sleeve Gastrectomy: a Prospective, Randomized, Single Blinded Clinical Trial
Brief Title: The Effect of Anesthetic Methods on Gastrointestinal Motility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, MD, Anesthesiology Specialist, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HandeBariatric
Record Dates: First submitted 2023-06-05; First posted 2023-07-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia; Total Intravenous Anesthesia
Keywords: gastric motility; laparoscopic sleeve gastrectomy; desflurane; propofol; remifentanil; peristalsis
MeSH Terms: interventions — Desflurane; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group inhalation (Active Comparator): Patients will receive desflurane as an inhalation anesthetic and remifentanil infusion for general anesthesia maintenance during the surgery. The doses of desflurane and remifentanil will be adjusted according to the Patient State Index (PSI) where the goal score is 25-50.
  Interventions: Drug: Desflurane; Drug: Remifentanil infusion; Other: Fresh gas
- Group tiva (Active Comparator): Patients will receive total intravenous anesthesia with an infusion of propofol and remifentanil for general anesthesia maintenance during the surgery. The infusion doses will be changed according to the Patient State Index (PSI) where the goal score is 25-50.
  Interventions: Drug: Remifentanil infusion; Other: Fresh gas; Drug: Propofol infusion

INTERVENTIONS:
Drug: Desflurane — In inhalation group, desflurane will be used for general anesthesia maintenance under the screening with Patient State Index (PSI) between a score of 25-50. Remifentanil infusion is used with desflurane with a dose of 0.05-2 mcg/ kg/ min according to PSI . Fresh gas flow is used 2 L/ min with a mixture of 50%- 50% oxygen and medical air in both groups.
  Other Names: suprane
  Arms: Group inhalation
Drug: Remifentanil infusion — Remifentanil infusion will be used with a dose of 0.05-2 mcg/ kg/ min under the screening with Patient State Index (PSI) between a score of 25-50 in both groups.
  Other Names: ultiva
Other: Fresh gas — Fresh gas flow will be used 2 L/ min with a mixture of 50%- 50% oxygen and medical air in both groups.
Drug: Propofol infusion — Propofol infusion will be used for general anesthesia maintenance with a dose of under the screening of Patient State Index (PSI) between a score of 25-50 in group tiva.
  Other Names: propofol 2%
  Arms: Group tiva

SUMMARY:
The goal of this randomized controlled single blinded study is to compare the effect of the type of anesthesia on gastrointestinal motility in patients scheduled for laparoscopic sleeve gastrectomy. The main question it aims to answer is how do inhalation anesthesia and total intravenous anesthesia effect the gastrointestinal peristalsis during anastomosis.

Participants will be American Society of Anesthesiology (ASA) physical status II and III, between 18- 60 ages.

Researchers will compare inhalation anesthesia where desflurane is used with total intravenous anesthesia to see if the gastrointestinal motility differs between the groups.

DETAILED DESCRIPTION:
Aim of this study is to evaluate the effect of two anesthetic methods on gastric motility during laparoscopic sleeve gastrectomy. Patients scheduled for laparoscopic sleeve gastrectomy with American Society of Anesthesiology (ASA) physical status II and III will enrolled into two groups. Computer based randomization will be used for the group selection. Patients will be monitored with standard monitorization (peripheral oxygen saturation, non-invasive blood pressure, 3-lead electrocardiography and patient state index (PSI)). Preoxygenation will be performed via a face mask with 6 L/min oxygen for 5 minutes. All patients will receive intravenous 2 mg/kg propofol, 0.25 mcg/kg/min remifentanil for anesthesia induction. Rocuronium bromide will be used intravenously with a dose of 0.6 mg/kg for muscle relaxation. Endotracheal intubation will be performed. In Group 1, inhalation anesthetic, desflurane and in Group 2, propofol infusion will be used with a 2 L/ min fresh gas flow as a mixture of 50 %- 50 % oxygen- medical air for maintenance of general anesthesia. Remifentanil infusion with a dose of 0.05-2 mcg/kg/min will be used in both groups during anesthesia maintenance. Anesthesia depth will be monitored with EEG monitorization where a score of 25-50 will be achieved in PSI . End-tidal carbon dioxide pressure will be kept between 35 and 45 mmHg. End-expiratory positive pressure will be set to 8 mmHg and intraabdominal pressure will be set to 12 mmHg. The surgeon will assess the gastric motility during anastomosis. The peristalsis during 1 minute period will be counted. 1 gram paracetamol and 1 mg/kg tramadol will be given intravenously for pain management. Sugammadex will be used for the reversal of neuromuscular blockade. Postoperative nause and vomiting, the time of first fart will be noted. Surgeon's satisfaction during anastomosis will be assessed with 5 points Likert Scale. Data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 ages
* ASA II-III
* Patients scheduled for elective laparoscopic sleeve gastrectomy
* Body mass index 35 kg m2 and over

Exclusion Criteria:

* Hepatic disease
* Kidney disease
* Congestive heart disease
* Diabetes mellitus
* Neurological deficit
* Psychiatric disease
* Pregnancy
* Delayed gastric empting
* Previous bariatric surgery
* Patient's refusal
* Open surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal motility | during surgery
  Gastrointestinal motility is the number of peristalsis during a one minute period. The surgeon will be asked to count the number of peristalsis during surgical anastomosis in a one minute period.

SECONDARY OUTCOMES:
Fart | up to 24 hours after surgery
  The time of first fart
Nause and vomiting | up to 24 hours after surgery
  Incidence of postoperative nause and vomiting
Satisfaction of surgeon | during surgery
  Ease of anastomosis and satisfaction of surgeon will be measured with 5 point Likert Scale as 1: very dissatisfied, 2:dissatisfied, 3: neither dissatisfied or satisfied, 4: satisfied, 5: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Halide H Şahinkaya, MD, Principal Investigator — Izmir Bozyaka Education and Research Hospital; Ahmet M Öztürk, MD, Study Chair — Izmir Bozyaka Education and Research Hospital; Çağlar Ayar, MD, Study Chair — Izmir Bozyaka Education and Research Hospital; Hüseyin Özkarakaş, MD, Study Chair — Izmir Bozyaka Education and Research Hospital; Bülent Çalık, Ass. Prof, Study Chair — Izmir Bozyaka Education and Research Hospital; Zeki T Tekgül, Ass. Prof., Study Chair — Izmir Bozyaka Education and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Bozyaka, Turkey (Türkiye)

REFERENCES:
- [Background] Akkurt BC, Temiz M, Inanoglu K, Aslan A, Turhanoglu S, Asfuroglu Z, Canbolant E. Comparison of recovery characteristics, postoperative nausea and vomiting, and gastrointestinal motility with total intravenous anesthesia with propofol versus inhalation anesthesia with desflurane for laparoscopic cholecystectomy: A randomized controlled study. Curr Ther Res Clin Exp. 2009 Apr;70(2):94-103. doi: 10.1016/j.curtheres.2009.04.002. PMID 24683221
- [Background] Liao Q, Wang MA, Ouyang W. [Effect of different anesthesias on gastrointestinal motility after laparoscopic cholecystectomy]. Hunan Yi Ke Da Xue Xue Bao. 2003 Feb 28;28(1):73-5. Chinese. PMID 12934407
- [Background] De Corte W, Delrue H, Vanfleteren LJ, Dutre PE, Pottel H, Devriendt DK, Van Rooy FH, D'Hondt M, Carlier S, Desmet MB. Randomized clinical trial on the influence of anaesthesia protocol on intestinal motility during laparoscopic surgery requiring small bowel anastomosis. Br J Surg. 2012 Nov;99(11):1524-9. doi: 10.1002/bjs.8883. Epub 2012 Sep 21. PMID 23001752